CLINICAL TRIAL: NCT03230331
Title: Long Term Study of Subthalamic Deep Brain Stimulation for Parkinson's Disease
Brief Title: Follow Up Study for Treatment of Parkinson's Disease With Subthalamic Deep Brain Stimulation
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Haiyan Zhou, Principal Investigator, Ruijin Hospital
Other Study IDs: FOGSTN
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STN DBS: Parkinson's disease (PD) patients who underwent deep brain stimulation (DBS) of the subthalamic nucleus (STN)
- CONTROL: Parkinson's disease (PD) patients received optimized medical treatment according to published evidence based guidelines

SUMMARY:
This study aims to evaluate the long term effect of deep brain stimulation in the the subthalamic nucleus (STN) in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* Disease duration longer than 15 years
* Had STN deep brain stimulation implant more than 10 years
* Available and willing to be followed-up according to study protocol

Exclusion Criteria:

* Patients with serious diseases such as tumor, sever liver or kidney dysfunction were not selected in the clinical trials
* Epilepsy
* Pregnant female
* History of severe neuropsychiatric disease
* Patients are taking part in other clinical trials in recent several months

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's Disease who underwent STN DBS for above 10 years or Patients with Parkinson's Disease whose disease duration longer than 15 years.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Changs in the score of Stand-Walk-Sit Test | above 10 years post surgery

SECONDARY OUTCOMES:
Change of the score in United Parkinson Disease Rating Scale (UPDRS) part III | above 10 years post surgery
UPDRS part I score | above 10 years post surgery
UPDRS part II score | above 10 years post surgery
UPDRS part IV score | above 10 years post surgery
39-Item Parkinson´s Disease Questionnaire (PDQ-39) score | above 10 years post surgery
Freezing of Gait Questionnaire (FOG-Q) score | above 10 years post surgery
Gait and Falls Questionnaire (GFQ) score | above 10 years post surgery
Mini-Mental State Examination (MMSE) score | above 10 years post surgery
Montreal Cognitive Assessment (MoCA) Beijing score Version | above 10 years post surgery
Frontal Assessment Battery (FAB) score | above 10 years post surgery
Hamilton Anxiety Scale (HAMA) score | above 10 years post surgery
Hamilton Depression Scale-17 (HAMD-17) score | above 10 years post surgery
Apathy Evaluation Scale score | above 10 years post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Zhou, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine; Dianyou Li, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine; Bomin Sun, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine; Wei Hu, Principal Investigator — University of Florida
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China